CLINICAL TRIAL: NCT03625518
Title: Mode of Induction in Fetal Growth Restriction and Its Affects on Fetal and Maternal Outcomes
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 0114-18
Record Dates: First submitted 2018-07-31; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Fetal Growth Retardation; Induction of Labor Affected Fetus / Newborn
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- prostaglandins (Active Comparator): vaginal prostaglandins insertion (PGE2) for cervical ripening and induction
  Interventions: Drug: prostaglandins E2
- intracervical balloon catheter with pitocin (Active Comparator): insertion of intra cervical balloon catheter combined with intravenous pitocin for ripening and induction of labor
  Interventions: Device: intracervical balloon catheter combined with pitocin

INTERVENTIONS:
Drug: prostaglandins E2 — insertion of vaginal PGE2 for up to 30 hours, up to two attempts for cervical ripening and induction
  Other Names: dinoprostone slow release pessary
  Arms: prostaglandins
Device: intracervical balloon catheter combined with pitocin — insertion of Foley catheter intra cervical and inflating the balloon with 50-60 cc of saline, with IV pitocin according to hospital protocol
  Arms: intracervical balloon catheter with pitocin

SUMMARY:
to compare methods of induction of labor in fetal growth restriction and its effect on maternal and neonatal outcome

DETAILED DESCRIPTION:
Intra uterine growth restriction (FGR) is a condition in which the fetus does not realize its growth potential in uterus. The excepted definitions of this condition are fetal weight estimation below the 10th percentile per gestational week. Severe growth restriction is defined as estimated weight below the 3rd percentile. It is well known that fetuses which are growth restricted are subjected to a higher degree of complications during pregnancy and delivery such as fetal distress, hypoxic damage, intra uterine fetal demise and complications in the neonatal period including prolonged NICU hospitalization, cerebral palsy, hypoxic ischemic encephalopathy and also long term affects such as neuro developmental complications.

Common practice in managing these cases is induction of labor at term around 37 weeks of gestations to prevent these complications as it established that during this time there is a substantial rise in pregnancy complications including fetal demise.

There are no clear guide lines how to induce labor in such cases and it is not known what is the safest and the most effective way to induce labor in these cases. Prior studies have found the rate of successful vaginal birth in these cases vary between 50 and 80%. There are a number of methods of labor induction and delivery available including the use of vaginal prostaglandins (PGE2) for cervical ripening, intracervical balloon catheter or planned cesarean. In most cases when aiming for vaginal delivery the choice is between ripening of the cervix with balloon catheter in combination with Pitocin or ripening with prostaglandins. It is not known which method is safer and more successful in growth restricted fetuses.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* fetal growth restriction defined as estimated fetal weight between the 3rd and 10th percentile per gestational age and are intended to deliver vaginally
* Gestational age between 36 and 42 weeks
* No known fetal anomalies

Exclusion Criteria:

* Fetal estimated weight below the 3rd percentile
* Known fetal anomalies
* Contraindications for vaginal delivery: breech presentation, abnormal Doppler flow velocimetry of fetal ductus venosus.
* Oligohydramnios defined as amniotic fluid index below 5 cm
* Contraindication to the use of prostaglandins
* Fetal distress requiring emergent cesarean section
* All other condition preventing vaginal delivery as decided by a senior physician

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 280 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
mode of delivery | immediate
  vaginal delivery, instrumental delivery or cesarean delivery

SECONDARY OUTCOMES:
composite neonatal outcome | 3 months after delivery
  apgar score at birth, umilical cord blood gases, neonatal intensive care unit hospitalization,Intra ventricular hemorrhage, periventricular leukomalacia, meconium aspiration syndrome, sepsis, convulsion, perinatal death, need for hypothermia treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Lis Maternity Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Figueras F, Gratacos E. Update on the diagnosis and classification of fetal growth restriction and proposal of a stage-based management protocol. Fetal Diagn Ther. 2014;36(2):86-98. doi: 10.1159/000357592. Epub 2014 Jan 23. PMID 24457811
- [Background] Baschat AA. Fetal growth restriction - from observation to intervention. J Perinat Med. 2010 May;38(3):239-46. doi: 10.1515/jpm.2010.041. PMID 20205623
- [Background] Walker DM, Marlow N. Neurocognitive outcome following fetal growth restriction. Arch Dis Child Fetal Neonatal Ed. 2008 Jul;93(4):F322-5. doi: 10.1136/adc.2007.120485. Epub 2008 Apr 1. PMID 18381841
- [Background] Boers KE, Vijgen SM, Bijlenga D, van der Post JA, Bekedam DJ, Kwee A, van der Salm PC, van Pampus MG, Spaanderman ME, de Boer K, Duvekot JJ, Bremer HA, Hasaart TH, Delemarre FM, Bloemenkamp KW, van Meir CA, Willekes C, Wijnen EJ, Rijken M, le Cessie S, Roumen FJ, Thornton JG, van Lith JM, Mol BW, Scherjon SA; DIGITAT study group. Induction versus expectant monitoring for intrauterine growth restriction at term: randomised equivalence trial (DIGITAT). BMJ. 2010 Dec 21;341:c7087. doi: 10.1136/bmj.c7087. PMID 21177352
- [Background] ACOG Practice bulletin no. 134: fetal growth restriction. Obstet Gynecol. 2013 May;121(5):1122-1133. doi: 10.1097/01.AOG.0000429658.85846.f9. PMID 23635765
- [Background] Horowitz KM, Feldman D. Fetal growth restriction: risk factors for unplanned primary cesarean delivery. J Matern Fetal Neonatal Med. 2015;28(18):2131-4. doi: 10.3109/14767058.2014.980807. Epub 2014 Nov 14. PMID 25354283
- [Background] Maslovitz S, Shenhav M, Levin I, Almog B, Ochshorn Y, Kupferminc M, Many A. Outcome of induced deliveries in growth-restricted fetuses: second thoughts about the vaginal option. Arch Gynecol Obstet. 2009 Feb;279(2):139-43. doi: 10.1007/s00404-008-0685-5. Epub 2008 May 28. PMID 18506461